CLINICAL TRIAL: NCT06707428
Title: Do Compression Stockings Used During Cesarean Sections Affect Intraoperative Hypotension and Nausea?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Seçil Yavaş, Ph.D. student in women's health and diseases nursing, TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ErciyesU-SBE-SY-01
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Intraoperative Hypotension
Keywords: hypotension; vasopressor; varicose veins
MeSH Terms: conditions — Hypotension; Varicose Veins | interventions — Stockings, Compression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression stocking using group (Experimental): Wearing varicose vein stockhing is a routine operation preparation
  Interventions: Other: compression stockings
- Control Group (No Intervention): Routine opreration preparation

INTERVENTIONS:
Other: compression stockings — compression stockings used during cesarean section
  Arms: Compression stocking using group

SUMMARY:
The present study aimed to determine the effects of compression stockings used during cesarean section on intraoperative hypotension.

DETAILED DESCRIPTION:
Cesarean section is among the most common surgeries in young and healthy individuals. Its frequency is increasing in our country and on a global scale. A total of 57% of all births in our country were performed by cesarean section between 2018 and 2023.

Spinal anesthesia is frequently used during cesarean sections with its advantages such as the patient being conscious, not having a risk of aspiration, not causing respiratory depression in the newborn, and the mother being able to breastfeed early. However, Spinal Anesthesia has complications such as hypotension and post-spinal headache, bradycardia and asystole, nausea, hypoventilation, total spinal block, urinary retention, spinal hematoma, back pain, infection, transient neurological symptoms, or cranial nerve paralysis. The present study aimed to determine the effects of compression stockings used during cesarean section on intraoperative hypotension.

ELIGIBILITY:
Inclusion Criteria:

37-38 weeks pregnant women

Exclusion Criteria:

* chronic disease
* women who developed complications during surgery
* women with multiple pregnancies
* women with pregnancies with known fetal anomalies

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 72 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
decrease in blood pressure | one year
  systolic blood pressure
decrease in blood pressure | one year
  diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Afşin Devlet Hastanesi, Afşin, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradhan, A., Das, T., Sraban, S., Pradhan, K., & Raut, K. (2016). Study the Hemodynamic changes after leg wrapping in elective cesarean section under spinal anesthesia. J Med Sci Clin Res, 4(11), 12-20.https://doi.org/10.18535/jmscr/v4i11.66
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Ferre F, Martin C, Bosch L, Kurrek M, Lairez O, Minville V. Control of Spinal Anesthesia-Induced Hypotension in Adults. Local Reg Anesth. 2020 Jun 3;13:39-46. doi: 10.2147/LRA.S240753. eCollection 2020. PMID 32581577
- [Background] Chang YJ, Liu CC, Huang YT, Wu JY, Hung KC, Liu PH, Lin CH, Lin YT, Chen IW, Lan KM. Assessing the Efficacy of Inferior Vena Cava Collapsibility Index for Predicting Hypotension after Central Neuraxial Block: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2023 Aug 31;13(17):2819. doi: 10.3390/diagnostics13172819. PMID 37685357
- [Background] Ağaçayak, E., Yavuz, M., Tunç, S. Y., Akın, G., Ertuğrul, S., Yıldırım, Z. B., & Gül, T. (2019). Comparison neonatal outcomes of elective cesareans performed with spinal or general anesthesia and normal births without anesthesia. Dicle Medical Journal , 46(2), 299-305.https://doi.org/10.5798/dicletip.574822
- [Background] Adatepe S. (2020). Comparison of neonatal outcomes of elective cesarean sections performed with spinal or general anesthesia and normal deliveries without anesthesia.Specialization Thesis. Tokat Gaziosmanpaşa University.
- [Result] Yu C, Gu J, Liao Z, Feng S. Prediction of spinal anesthesia-induced hypotension during elective cesarean section: a systematic review of prospective observational studies. Int J Obstet Anesth. 2021 Aug;47:103175. doi: 10.1016/j.ijoa.2021.103175. Epub 2021 May 1. PMID 34034957
- [Result] Ebrahim Elgzar WT, Ebrahim Said H, Ebrahim HA. Effect of lower leg compression during cesarean section on post-spinal hypotension and neonatal hemodynamic parameters: nonrandomized controlled clinical trial. Int J Nurs Sci. 2019 Jun 10;6(3):252-258. doi: 10.1016/j.ijnss.2019.06.003. eCollection 2019 Jul 10. PMID 31508443
- [Result] Ulgu MM, Birinci S, Altun Ensari T, Gozukara MG. Cesarean section rates in Turkey 2018-2023: Overview of national data by using Robson ten group classification system. Turk J Obstet Gynecol. 2023 Sep 4;20(3):191-198. doi: 10.4274/tjod.galenos.2023.68235. PMID 37667479
- [Result] Mohamed AI, Elazhary RA, Abdelhady RM, Abd-ElSadek BR, Said KM. Utilization of lower leg compression technique for reducing spinal induced hypotension, and related risks for mothers and neonates during cesarean delivery. J Nurs Educ Pract 2016;6(7):11e8. https://doi.org/10.5430/jnep.v6n7p11
- [Result] Mohamad A., Rama B., Farshid G., Kourosh F., Reza A. (2020). A randomized double-blind clinical trial evaluating the effect of Elastic Stocking on Hemodynamic Changes and dose use of ephedrine for elective cesarean surgery under spinal anesthesia. International Journal of Surgery Open, 27, 58-63, https://doi.org/10.1016/j.ijso.2020.10.019
- [Result] Wan L, Shen PY, Zhang SX, Wang LZ. Leg Compression Versus Control for Prevention of Spinal Anesthesia Induced Hypotension in Elective Cesarean Delivery: A Meta-Analysis of Randomized Controlled Trials. J Perianesth Nurs. 2022 Aug;37(4):501-508. doi: 10.1016/j.jopan.2021.10.011. Epub 2022 Mar 4. PMID 35256251
- [Result] Yao HQ, Huang JY, Dong YF, Sun XX, Wang LZ. Effect of pneumatic leg compression on phenylephrine dose for hypotension prophylaxis via variable rate infusion at cesarean delivery: an unblinded randomized controlled trial. Int J Obstet Anesth. 2024 Nov;60:104218. doi: 10.1016/j.ijoa.2024.104218. Epub 2024 Jun 11. PMID 38925990
- [Result] Hasanin A, Aiyad A, Elsakka A, Kamel A, Fouad R, Osman M, Mokhtar A, Refaat S, Hassabelnaby Y. Leg elevation decreases the incidence of post-spinal hypotension in cesarean section: a randomized controlled trial. BMC Anesthesiol. 2017 Apr 24;17(1):60. doi: 10.1186/s12871-017-0349-8. PMID 28438121